CLINICAL TRIAL: NCT01980732
Title: 68Ga DOTA-TATE PET/CT in the Evaluation of Patients With Somatostatin Receptor Positive Tumors
Brief Title: 68Ga DOTA-TATE PET/CT in Somatostatin Receptor Positive Tumors
Status: No longer available | Type: Expanded Access
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Assistant Professor of Radiology - Nuclear Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: NET0017; 26988
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Carcinoid Tumors; Islet Cell (Pancreatic NET); Other Neuroendocrine Tumors
MeSH Terms: conditions — Carcinoid Tumor; Adenoma, Islet Cell | interventions — gallium Ga 68 dotatate

INTERVENTIONS:
Drug: 68Ga-DOTA TATE — Patients with somatostatin receptor positive tumors will be evaluated with 68Ga-DOTA TATE PET/CT in addition to conventional imaging.

SUMMARY:
The primary objective of the study is to evaluate 68Ga-DOTA TATE PET/CT for staging and monitoring response to chemotherapy in patients with carcinoid, neuroendocrine tumors, medullary thyroid cancer and other cancers expressing somatostatin receptors.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years-old at the time of radiotracer administration
* Provides written informed consent
* Known diagnosis of NET or suspected SSTR positive tumors by 111In-Octreotide scan, 18FDG-PET, or MRI of the abdomen when clinically indicated
* Karnofsky score greater than 50 or ECOG Performance Status 0-2
* Women of childbearing age must have a negative pregnancy test at screening/baseline
* Able to remain still for duration of each imaging procedure (about one hour)

Exclusion Criteria:

* Less than 18 years-old at the time of radiotracer administration
* Pregnant or nursing
* Serum creatinine >3.0 mg/dL
* Hepatic enzyme levels more than 5 times upper limit of normal.
* Use of any other investigational product or device within 30 days prior to dosing, or known requirement for any other investigational agent prior to completion of all scheduled study assessments.
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States